CLINICAL TRIAL: NCT02858362
Title: Phaseout DMD: A Phase 2 Clinical Study to Assess the Activity and Safety of Utrophin Modulation With Ezutromid in Ambulatory Paediatric Male Subjects With Duchenne Muscular Dystrophy (SMT C11005)
Brief Title: Proof of Concept Study to Assess Activity and Safety of SMT C1100 (Ezutromid) in Boys With Duchenne Muscular Dystrophy (DMD)
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: The study was terminated due to lack of efficacy in Cohorts 1 and 2.
Sponsor: Summit Therapeutics (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: SMT C11005; 2015-004333-27 (EudraCT Number)
Record Dates: First submitted 2016-07-27; First posted 2016-08-08 (Estimated); Results first posted 2020-01-02 (Actual); Last update posted 2020-01-02 (Actual); Status verified 2019-12

CONDITIONS: Duchenne Muscular Dystrophy
Keywords: DMD; Muscular Dystrophy; Utrophin; Duchenne; PhaseOut DMD
MeSH Terms: conditions — Muscular Dystrophy, Duchenne; Muscular Dystrophies | interventions — ezutromid; SMT C1100

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- Cohort 1: SMT C1100 Formulation 1 (Experimental): Participants received 2.5 g SMT C1100 formulation 1 orally twice-daily for at least 48 weeks.
  Interventions: Drug: Ezutromid
- Cohort 2: SMT C1100 Formulation 2 (Experimental): Participants received 1 g SMT C1100 formulation 2 orally twice-daily for at least 48 weeks.
  Interventions: Drug: Ezutromid
- Cohort 3: SMT C1100 Formulation 1 (Experimental): Participants in this cohort had previously received SMT C1100, but were not eligible for Cohorts 1 or 2. Participants received 2.5 g SMT C1100 formulation 1 orally twice-daily for at least 48 weeks.
  Interventions: Drug: Ezutromid

INTERVENTIONS:
Drug: Ezutromid — Administered orally.
  Other Names: SMT C1100

SUMMARY:
To Assess the Activity and Safety of SMT C1100 (Ezutromid) in Paediatric Male Participants with Duchenne Muscular Dystrophy (DMD).

DETAILED DESCRIPTION:
This is a Phase 2, open label, study to assess the activity and safety of utrophin modulation with SMT C1100 (ezutromid) administered twice-daily orally in ambulatory paediatric male participants with DMD.

This study will be conducted in a multi-centre setting in both the United Kingdom and the United States of America and comprises of a Screening and Baseline Phase of up to 28 days, a 48-week open label Treatment Phase, and either a 30-day Safety Follow up Phase or an optional extension phase where study treatment is provided until discontinuation of the program or regulatory approvals as applicable.

ELIGIBILITY:
Inclusion Criteria:

* Be able to provide written informed consent/assent as per local requirements.
* Be male.
* Have phenotypic evidence of dystrophinopathy based on the onset of characteristic clinical symptoms or signs (e.g., proximal muscle weakness, waddling gait, and Gowers' manoeuvre), an elevated serum creatinine kinase level, and ongoing difficulty with walking.
* Have prior confirmation of the duchenne muscular dystrophy (DMD) diagnosis through:

Documentation of the presence of a mutation in the dystrophin gene as determined by gene sequencing from a laboratory certified by the College of American Pathologists, the Clinical Laboratory Improvement Act/Amendment or an equivalent organisation or documentation of the absence of dystrophin in the muscle (via biopsy).

* Be able to undergo MRI examination.
* Participants must have used stable systemic corticosteroids (prednisone, prednisolone or deflazacort) for a minimum of 6 months immediately prior to the start of the Treatment Phase, with no significant change in dosage or dosing regimen (not related to body weight change) and a reasonable expectation that dosage and dosing regimen will not change significantly for the duration of the study.
* Confirmed screening laboratory values within the central laboratory ranges (haematology, renal and serum electrolyte parameters and serum chemistry parameters) or considered not clinically significant in the opinion of the Investigator. Variations in specific parameters expected in a DMD population classed by the Investigator as not clinically significant will not exclude the participant.
* Be willing and able to comply with scheduled visits, drug administration plan, study procedures, laboratory tests and study restrictions.

Cohort 1 and 2 Specific Inclusion Criteria:

* Be aged ≥5 years to <10 years of age (from 5th birthday to 10th birthday).
* Be willing and able to comply with 2 muscle biopsy procedures.
* Have the ability to walk at least 300 meters unassisted during the screening 6 minute walk distance (6MWD) and be below the protocol-specified threshold for 80%-predicted 6MWD.
* Have results of 2 6MWD by Baseline determined as valid. The results of the second 6MWD (baseline) must be within 20% of the first 6MWD (screening).
* Have cardiac echocardiogram (ECHO) measurements showing an ejection fraction of ≥55% and fractional shortening of ≥28%.

Cohort 3 Specific Inclusion Criteria:

* Have taken part in a prior SMT C1100 study.

Exclusion Criteria:

* Have physical exam findings that in the Investigator's opinion should be exclusionary e.g., lower limb injury that may affect 6MWD performance.
* Have any change (initiation, change in type of drug, dose modification, schedule modification, interruption, discontinuation or reinitiation) in prophylaxis/treatment for congestive heart failure (CHF) within 3 months prior to the start of study treatment.
* Have uncontrolled clinical symptoms and signs of CHF (American College of Cardiology/American Heart Association Stage C or Stage D).
* Have abnormal glutamate dehydrogenase (GLDH) at baseline (>1.5 x upper limit of normal [ULN]).
* Have abnormal coagulation times at baseline (>1.5 x ULN).
* Have an abnormal electrocardiograms (ECG).
* Use herbal supplements and be unwilling to stop these for the duration of the study.
* Have been exposed to another investigational drug or DMD interventional agent within 3 months prior to start of the Treatment Phase. Prior exposure to SMT C1100 or participation in an approved deflazacort access program within this period would not exclude the participant (provided they have been on stable treatment for 6 months).
* Have a history of major surgical procedure within 12 weeks prior to the start of the Treatment Phase (Week 1).
* Be undertaking ongoing immunosuppressive therapy (other than corticosteroids).
* Require daytime ventilator assistance.
* Have a prior or ongoing medical condition, medical history, ECG findings, or laboratory abnormality that, in the Investigator's opinion, could adversely affect the safety of the participant, makes it unlikely that the course of treatment or follow-up would be completed, or could impair the assessment of study results.
* Be dairy or lactose intolerant or have any other dietary restrictions that might interfere with the conduct of the study.
* Be a smoker, use other tobacco or nicotine products or be exposed to daily passive smoking (including parent/legal guardian, siblings) so as to minimise environmental factors causing CYP1A induction.
* Be using an approved DMD medication or anticipates using one during the duration of the study. Participants who are taking part in the FOR-DMD and ACCESS DMD studies will be allowed to take part.
* Be using an inducer of CYP1A1 or CYP1A2.
* Be using a substrate of CYP2B6.
* All prescription, over the counter, and herbal products that are known CYP2B6 sensitive substrates will be excluded 14 days prior to study conduct (beginning at screening) through 14 days after study conduct completion. Please note, this is not an exhaustive list of CYP2B6 substrates and a discussion with the Medical Monitor may be warranted.
* Be using drugs that have serotonergic, norepinephrinergic or dopaminergic activity, or treatments used in attention deficit hyperactivity disorder.
* Use of substrates of BRCP.

Cohort 1 and 2 Specific Exclusion Criteria:

* Use beta blockers (however, if during the course of the study they are clinically indicated they can be initiated).

Cohort 1 and 3 Specific Exclusion Criteria:

* Have a known hypersensitivity to any of the ingredients or excipients of the investigational medicinal product: Poloxamer 188, Methylparaben, Propylparaben, Hydroxypropylmethyl cellulose, Glycerol, Non-crystallising sorbitol [70%], Xanthan gum, Strawberry cream flavour [PHS-132963].

Cohort 2 Specific Exclusion Criteria:

* Have a known hypersensitivity to any of the ingredients or excipients of the investigational medicinal product: hypromellose acetate succinate.

Min Age: 5 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 43 (Actual)
Dates: Start 2016-06 (Actual); Primary Completion 2018-04-11 (Actual); Study Completion 2018-09-11 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Medical Monitor, Study Director — Summit (Oxford) Limited
Locations (16):
- United States (9):
  - UCLA-David Geffen School of Medicine, Los Angeles, California
  - Children's Hosptial of Colorado, Aurora, Colorado
  - Nemours Children's Clinic, Orlando, Florida
  - Boston Children's Hospital, Boston, Massachusetts
  - Cincinnati Children's Hospital Medical Center, Cincinnati, Ohio
  - Oregon Health and Science University, Portland, Oregon
  - Children's Hospital of Philadelphia, Philadelphia, Pennsylvania
  - Vanderbilt University Medical Center, Nashville, Tennessee
  - University of Utah Hospital and Clinics, Salt Lake City, Utah
- United Kingdom (7):
  - Heart of England NHS Foundation Trust - Heartlands Hospital, Birmingham
  - Bristol Children's Hospital, Bristol
  - Addenbrooke's Hospital, Cambridge
  - Alder Hey Children's NHS Foundation Trust, Liverpool
  - Great Ormond Street Hospital for Children NHS Foundation Trust, London
  - Royal Manchester Children's Hospital - Central Manchester University Hospitals NHS Foundation Trust, Manchester
  - The Freeman Hospital, Newcastle Upon Tyne Hospitals, Newcastle

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants were enrolled in 16 sites across the United Kingdom (UK) and United States (US) between the dates of 16 June 2016 (First Patient In) and 11 September 2018 (Last Patient Out). Cohort 1 was conducted in the UK and US, Cohort 2 was conducted in the US only, and Cohort 3 was conducted in the UK only.
Period: Overall Study
Arm/Group | Cohort 1: SMT C1100 Formulation 1 | Cohort 2: SMT C1100 Formulation 2 | Cohort 3: SMT C1100 Formulation 1
Started | 30 | 10 | 3
Did Not Enter Extension Phase (Completed the study (Week 48 treatment visit) but did not enter the optional extension phase.) | 1 | 2 | 0
Completed | 28 | 9 | 0
Not Completed | 2 | 1 | 3
Not completed — Protocol Violation | 0 | 1 | 0
Not completed — Withdrawal by Subject | 1 | 0 | 0
Not completed — Early Study Termination | 0 | 0 | 3
Not completed — Lost to Follow-up | 1 | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Cohort 1: SMT C1100 Formulation 1 | Cohort 2: SMT C1100 Formulation 2 | Cohort 3: SMT C1100 Formulation 1 | Total
Number analyzed (Participants) | 30 | 10 | 3 | 43
Age, Customized [Count of Participants; unit: Participants]
  Children (2-11 years) | 30 | 10 | 1 | 41
  Adolescents (12-17 years) | 0 | 0 | 2 | 2
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0 | 0 | 0 | 0
  Male | 30 | 10 | 3 | 43
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 1 | 2 | 0 | 3
  Not Hispanic or Latino | 29 | 8 | 3 | 40
  Unknown or Not Reported | 0 | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0
  Asian | 1 | 1 | 0 | 2
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0
  Black or African American | 0 | 0 | 0 | 0
  White | 26 | 9 | 3 | 38
  More than one race | 2 | 0 | 0 | 2
  Unknown or Not Reported | 1 | 0 | 0 | 1
Magnetic Resonance Spectroscopy (MRS) Fat Fraction (FF) Vastus Lateralis [Mean (Standard Deviation); unit: Percentage of fat in the muscle] — Population: Efficacy measurements were planned and performed for Cohorts 1 and 2 only. One participant in Cohort 1 did not have analyzable results for MRS FF vastus lateralis at the baseline visit.
  Percentage of fat in the muscle
    number analyzed (Participants) | 29 | 10 | 0 | 39
    (all) | 13.78 (13.317) | 18.36 (13.664) |  | 14.95 (13.379)
Magnetic Resonance Spectroscopy (MRS) Fat Fraction (FF) Soleus [Mean (Standard Deviation); unit: Percentage of fat in the muscle] — Population: Efficacy measurements were planned and performed for Cohorts 1 and 2 only.
  Percentage of fat in the muscle
    number analyzed (Participants) | 30 | 10 | 0 | 40
    (all) | 8.57 (8.240) | 10.79 (9.996) |  | 9.12 (8.631)
Magnetic Resonance Spectroscopy (MRS) Water Transverse Relaxation Time (WTRT) Vastus Lateralis [Mean (Standard Deviation); unit: Milliseconds] — Population: Efficacy measurements were planned and performed for Cohorts 1 and 2 only. One participant in Cohort 1 did not have analyzable results for MRS WTRT vastus lateralis at the baseline visit.
  Milliseconds
    number analyzed (Participants) | 29 | 10 | 0 | 39
    (all) | 32.24 (1.980) | 32.17 (2.146) |  | 32.23 (1.995)
Magnetic Resonance Spectroscopy (MRS) Water Transverse Relaxation Time (WTRT) Soleus [Mean (Standard Deviation); unit: Milliseconds] — Population: Efficacy measurements were planned and performed for Cohorts 1 and 2 only.
  Milliseconds
    number analyzed (Participants) | 30 | 10 | 0 | 40
    (all) | 31.88 (1.936) | 31.87 (1.988) |  | 31.88 (1.923)
Development Heavy Chain Myosin (MHCd) Expression in Muscle Fibres [Mean (Standard Deviation); unit: Percent of muscle fibres expressing MHCd] — Population: Efficacy measurements were planned and performed for Cohorts 1 and 2 only. One participant in Cohort 1 did not have analyzable results for MHCd expression at the baseline visit.
  Percent of muscle fibres expressing MHCd
    number analyzed (Participants) | 29 | 10 | 0 | 39
    (all) | 12.185 (3.8454) | 11.587 (4.1344) |  | 12.032 (3.8748)
Muscle Fibre Diameter [Mean (Standard Deviation); unit: Micrometer] — Population: Efficacy measurements were planned and performed for Cohorts 1 and 2 only. One participant in Cohort 1 did not have analyzable results for muscle fibre diameter at the baseline visit.
  Micrometer
    number analyzed (Participants) | 29 | 10 | 0 | 39
    (all) | 43.662 (5.3837) | 42.086 (6.1878) |  | 43.258 (5.5598)
Utrophin Intensity [Mean (Standard Deviation); unit: Arbitrary Units] — Utrophin intensity is measured in arbitrary units (0-1) with higher scores representing higher utrophin expression. Population: Efficacy measurements were planned and performed for Cohorts 1 and 2 only. One participant in Cohort 2 did not have analyzable results for utrophin expression at the baseline visit.
  Arbitrary Units
    number analyzed (Participants) | 30 | 9 | 0 | 39
    (all) | 0.368 (0.0480) | 0.349 (0.0507) |  | 0.364 (0.0486)

OUTCOME MEASURES:

1. Primary Outcome: Change From Baseline in Magnetic Resonance Spectroscopy (MRS) Fat Fraction (FF) for Leg Muscles
Description: MRS FF was analysed for vastus lateralis and soleus leg muscles. The endpoints were measured for Cohorts 1 and 2 only. Results for Cohorts 1 and 2 are pooled as specified in the protocol.
Time Frame: Baseline, Week 12, Week 24, Week 36 and Week 48
Population: All participants who received at least one dose of study medication and had at least one assessment of the endpoint (which could be their baseline assessment).
Measure: Mean (95% Confidence Interval); unit: Percentage of fat in the muscle
Groups:
- Cohorts 1 and 2: SMT C1100: Cohort 1 participants received 2.5 g SMT C1100 formulation 1 orally twice-daily for at least 48 weeks. Cohort 2 participants received 1 g SMT C1100 formulation 2 orally twice-daily for at least 48 weeks.
Arm/Group | Cohorts 1 and 2: SMT C1100
Number analyzed (Participants) | 40
Percentage of fat in the muscle
  Vastus Lateralis: Week 12 Change from Baseline: number analyzed (Participants) | 39
  Vastus Lateralis: Week 12 Change from Baseline | 1.779 [0.939 to 2.620]
  Vastus Lateralis: Week 24 Change from Baseline: number analyzed (Participants) | 36
  Vastus Lateralis: Week 24 Change from Baseline | 3.914 [2.695 to 5.132]
  Vastus Lateralis: Week 36 Change from Baseline: number analyzed (Participants) | 37
  Vastus Lateralis: Week 36 Change from Baseline | 5.238 [3.563 to 6.913]
  Vastus Lateralis: Week 48 Change from Baseline: number analyzed (Participants) | 36
  Vastus Lateralis: Week 48 Change from Baseline | 7.142 [4.866 to 9.417]
  Soleus: Week 12 Change from Baseline | 0.615 [0.068 to 1.162]
  Soleus: Week 24 Change from Baseline: number analyzed (Participants) | 38
  Soleus: Week 24 Change from Baseline | 1.108 [0.350 to 1.865]
  Soleus: Week 36 Change from Baseline: number analyzed (Participants) | 38
  Soleus: Week 36 Change from Baseline | 2.384 [1.287 to 3.481]
  Soleus: Week 48 Change from Baseline: number analyzed (Participants) | 37
  Soleus: Week 48 Change from Baseline | 2.584 [1.258 to 3.909]

2. Primary Outcome: Change From Baseline for Magnetic Resonance Spectroscopy (MRS) Water Transverse Relaxation Time (WTRT) for Leg Muscles
Description: MRS WTRT was analysed for the vastus lateralis and soleus leg muscles. The endpoints were measured for Cohorts 1 and 2 only. Results for Cohorts 1 and 2 are pooled as specified in the protocol.
Time Frame: Baseline, Week 12, Week 24, Week 36 and Week 48
Population: as for outcome 1
Measure: Mean (95% Confidence Interval); unit: Milliseconds
Arm/Group | Cohorts 1 and 2: SMT C1100
Number analyzed (Participants) | 40
Milliseconds
  Vastus Lateralis: Week 12 Change from Baseline: number analyzed (Participants) | 39
  Vastus Lateralis: Week 12 Change from Baseline | -0.559 [-1.190 to 0.072]
  Vastus Lateralis: Week 24 Change from Baseline: number analyzed (Participants) | 36
  Vastus Lateralis: Week 24 Change from Baseline | -0.486 [-1.193 to 0.221]
  Vastus Lateralis: Week 36 Change from Baseline: number analyzed (Participants) | 37
  Vastus Lateralis: Week 36 Change from Baseline | -0.849 [-1.454 to -0.244]
  Vastus Lateralis: Week 48 Change from Baseline: number analyzed (Participants) | 36
  Vastus Lateralis: Week 48 Change from Baseline | -0.822 [-1.673 to 0.028]
  Soleus: Week 12 Change from Baseline | -0.655 [-1.209 to -0.101]
  Soleus: Week 24 Change from Baseline: number analyzed (Participants) | 38
  Soleus: Week 24 Change from Baseline | -0.861 [-1.440 to -0.281]
  Soleus: Week 36 Change from Baseline: number analyzed (Participants) | 38
  Soleus: Week 36 Change from Baseline | -0.447 [-1.085 to 0.190]
  Soleus: Week 48 Change from Baseline: number analyzed (Participants) | 37
  Soleus: Week 48 Change from Baseline | -0.119 [-0.747 to 0.509]

3. Primary Outcome: Observed Trough Plasma Concentration (Ctrough) for SMT C1100, Dihydrodiol 1 (DHD1) and Dihydrodiol III (DHD 3)
Description: Pharmacokinetic analysis is presented by cohort due to the use of different formulations. The median pre-dose concentration was derived for each participant and then summarized across participants.
Time Frame: Pre-dose at Weeks 1, 4, 8, 12, 24, 36 and 48
Population: All participants in Cohorts 1 or 2 who received at least one dose of study medication and had at least one concentration measurement (which could be below the limit of quantification). No evaluable data was collected from Cohort 3 participants due to early study termination.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ng/mL
Arm/Group | Cohort 1: SMT C1100 Formulation 1 | Cohort 2: SMT C1100 Formulation 2
Number analyzed (Participants) | 30 | 10
ng/mL
  SMT C1100 | 17 (140) | 80 (83.1)
  DHD 1 | 155 (61) | 365 (55)
  DHD 3 | 484 (67) | 1206 (68)

4. Primary Outcome: Simulated Maximum Plasma Concentration (Cmax) for SMT C1100, Dihydrodiol 1 (DHD1) and Dihydrodiol III (DHD 3)
Description: Pharmacokinetic analysis is presented by cohort due to the use of different formulations.
Time Frame: Pre-dose and 3 to 10 hours post-dose at Weeks 1, 4, 8, 12, 24, 36 and 48
Population: as for outcome 3
Measure: Geometric Mean (Full Range); unit: ng/mL
Arm/Group | Cohort 1: SMT C1100 Formulation 1 | Cohort 2: SMT C1100 Formulation 2
Number analyzed (Participants) | 30 | 10
ng/mL
  SMT C1100 | 135 [97 to 185] | 415 [303 to 640]
  DHD 1 | 1897 [1690 to 2158] | 2829 [2597 to 3072]
  DHD 3 | 3162 [2392 to 4053] | 4652 [3802 to 6116]

5. Primary Outcome: Simulated Average Plasma Concentration (Cav) for SMT C1100, Dihydrodiol 1 (DHD1) and Dihydrodiol III (DHD 3)
Description: Pharmacokinetic analysis is presented by cohort due to the use of different formulations.
Time Frame: Pre-dose and 3 to 10 hours post-dose at Weeks 1, 4, 8, 12, 24, 36 and 48
Population: as for outcome 3
Measure: Geometric Mean (Full Range); unit: ng/mL
Arm/Group | Cohort 1: SMT C1100 Formulation 1 | Cohort 2: SMT C1100 Formulation 2
Number analyzed (Participants) | 30 | 10
ng/mL
  SMT C1100 | 54 [37 to 82] | 163 [114 to 272]
  DHD 1 | 742 [685 to 836] | 1109 [1028 to 1217]
  DHD 3 | 1359 [972 to 1790] | 2211 [1707 to 3066]

6. Primary Outcome: Number of Participants Reporting One or More Treatment-Emergent Adverse Events (TEAEs)
Description: An adverse event is defined as any untoward medical occurrence in a patient or clinical investigation participant administered a pharmaceutical product and which does not necessarily have a causal relationship with this treatment. A TEAE is defined as any event not present before exposure to study drug or any event already present that worsens in either intensity or frequency after exposure to study drug.
Time Frame: Day 1 to a maximum of Week 96
Population: All participants who received at least one dose of study medication.
Measure: Count of Participants; unit: Participants
Arm/Group | Cohort 1: SMT C1100 Formulation 1 | Cohort 2: SMT C1100 Formulation 2 | Cohort 3: SMT C1100 Formulation 1
Number analyzed (Participants) | 30 | 10 | 3
Participants | 30 | 10 | 3

7. Secondary Outcome: Change From Baseline in Utrophin Intensity
Description: A maximum of two muscle biopsies were taken, one at baseline and the other at Week 24 or Week 48. Utrophin intensity was analyzed using a semiautomated quantitative assay on the biopsy samples. A positive change from baseline represents an increase in utrophin expression, no change from baseline represents maintenance of utrophin expression and a negative change from baseline represents a reduction in utrophin expression. The endpoint was measured for Cohorts 1 and 2 only. Results for Cohorts 1 and 2 are pooled as specified in the protocol.
Time Frame: Baseline, Week 24 and Week 48
Population: All participants who received at least one dose of study medication and had at least one assessment of the endpoint (which could be their baseline assessment). For the summaries of changes from baseline only those participants in this population who had measurements at both baseline and the relevant post-baseline visit were included.
Measure: Mean (Standard Deviation); unit: Arbitrary units
Arm/Group | Cohorts 1 and 2: SMT C1100
Number analyzed (Participants) | 37
Arbitrary units
  Change from baseline at Week 24: number analyzed (Participants) | 22
  Change from baseline at Week 24 | 0.0232 (0.0601)
  Change from baseline at Week 48: number analyzed (Participants) | 15
  Change from baseline at Week 48 | 0.0114 (0.0574)
Statistical Analysis 1: Comparison: Cohorts 1 and 2: SMT C1100; Week 24 Change from Baseline; Test type: Other — Difference in least square means. All 23 participants in the population were included in the statistical analysis; Mean Difference (Final Values) = 0.023, 95% CI 2-sided [-0.002 to 0.048]
Statistical Analysis 2: Comparison: Cohorts 1 and 2: SMT C1100; Week 48 Change from Baseline; Test type: Other — Difference in least square means. All 16 participants in the population were included in the statistical analysis; Mean Difference (Final Values) = 0.006, 95% CI 2-sided [-0.03 to 0.042]

8. Secondary Outcome: Change From Baseline in Developmental Heavy Chain Myosin (MHCd) Expression
Description: A maximum of two muscle biopsies were taken, one at baseline and the other at Week 24 or Week 48. MHCd expression was analyzed using a semiautomated quantitative assay on the biopsy samples. A positive change from baseline represents an increase in MHCd expression, no change from baseline represents maintenance of MHCd expression and a negative change from baseline represents a reduction in MHCd expression. The endpoint was measured for Cohorts 1 and 2 only. Results for Cohorts 1 and 2 are pooled as specified in the protocol.
Time Frame: Baseline, Week 24 and Week 48
Population: as for outcome 7
Measure: Mean (Standard Deviation); unit: Percent of muscle fibres expressing MHCd
Arm/Group | Cohorts 1 and 2: SMT C1100
Number analyzed (Participants) | 38
Percent of muscle fibres expressing MHCd
  Change from baseline at Week 24: number analyzed (Participants) | 22
  Change from baseline at Week 24 | -2.3166 (3.9180)
  Change from baseline at Week 48: number analyzed (Participants) | 16
  Change from baseline at Week 48 | 1.2248 (4.2596)
Statistical Analysis 1: Comparison: Cohorts 1 and 2: SMT C1100; Week 24 Change from Baseline; Test type: Other — Difference in least square means. All 24 participants in the population were included in the statistical analysis; Mean Difference (Final Values) = -2.611, 95% CI 2-sided [-4.324 to -0.898]
Statistical Analysis 2: Comparison: Cohorts 1 and 2: SMT C1100; Week 48 Change from Baseline; Test type: Other — Difference in least square means. All 16 participants in the population were included in the statistical analysis; Mean Difference (Final Values) = 1.166, 95% CI 2-sided [-1.103 to 3.435]

9. Secondary Outcome: Change From Baseline in Muscle Fibre Diameter
Description: A maximum of two muscle biopsies were taken, one at baseline and the other at Week 24 or Week 48. Muscle fibre diameter was analyzed using a semiautomated quantitative assay on the biopsy samples. The endpoint was measured for Cohorts 1 and 2 only. Results for Cohorts 1 and 2 are pooled as specified in the protocol.
Time Frame: Baseline, Week 24 and Week 48
Population: as for outcome 7
Measure: Mean (Standard Deviation); unit: Micrometers (μm)
Arm/Group | Cohorts 1 and 2: SMT C1100
Number analyzed (Participants) | 38
Micrometers (μm)
  Change from baseline at Week 24: number analyzed (Participants) | 22
  Change from baseline at Week 24 | -1.9205 (4.7250)
  Change from baseline at Week 48: number analyzed (Participants) | 16
  Change from baseline at Week 48 | 2.0636 (4.1267)
Statistical Analysis 1: Comparison: Cohorts 1 and 2: SMT C1100; Week 24 Change from Baseline; Test type: Other — Difference in least square means. All 24 participants in the population were included in the statistical analysis; Mean Difference (Final Values) = -1.837, 95% CI 2-sided [-3.989 to 0.315]
Statistical Analysis 2: Comparison: Cohorts 1 and 2: SMT C1100; Week 48 Change from Baseline; Test type: Other — Difference in least square means. All 16 participants in the population were included in the statistical analysis; Mean Difference (Final Values) = 2.21, 95% CI 2-sided [0.096 to 4.324]

10. Secondary Outcome: Change From Baseline in Forced Expiratory Volume in 1 Second (FEV1)
Description: Results for Cohorts 1, 2 and 3 are pooled as specified in the protocol.
Time Frame: Baseline, Week 12, Week 24, Week 36 and Week 48
Population: All participants who received at least one dose of study medication. No evaluable data was collected from Cohort 3 participants due to early study termination.
Measure: Mean (Standard Deviation); unit: Percentage of FEV1
Groups:
- Cohorts 1, 2 and 3: SMT C1100: Cohorts 1 and 3 participants received 2.5 g SMT C1100 formulation 1 orally twice-daily for at least 48 weeks. Cohort 2 participants received 1 g SMT C1100 formulation 2 orally twice-daily for at least 48 weeks.
Arm/Group | Cohorts 1, 2 and 3: SMT C1100
Number analyzed (Participants) | 38
Percentage of FEV1
  Week 12 Change from Baseline | -3.4 (20.86)
  Week 24 Change from Baseline: number analyzed (Participants) | 37
  Week 24 Change from Baseline | -2.5 (24.88)
  Week 36 Change from Baseline: number analyzed (Participants) | 36
  Week 36 Change from Baseline | -7.3 (24.26)
  Week 48 Change from Baseline: number analyzed (Participants) | 33
  Week 48 Change from Baseline | 2.0 (18.31)

11. Secondary Outcome: Change From Baseline in Forced Vital Capacity (FVC)
Description: Results for Cohorts 1, 2 and 3 are pooled as specified in the protocol.
Time Frame: Baseline, Week 12, Week 24, Week 36 and Week 48
Population: as for outcome 10
Measure: Mean (Standard Deviation); unit: Percentage of FVC
Arm/Group | Cohorts 1, 2 and 3: SMT C1100
Number analyzed (Participants) | 39
Percentage of FVC
  Week 12 Change from Baseline | -4.0 (16.31)
  Week 24 Change from Baseline: number analyzed (Participants) | 38
  Week 24 Change from Baseline | 1.1 (16.75)
  Week 36 Change from Baseline: number analyzed (Participants) | 37
  Week 36 Change from Baseline | -3.4 (18.39)
  Week 48 Change from Baseline: number analyzed (Participants) | 35
  Week 48 Change from Baseline | 1.1 (16.29)

12. Secondary Outcome: Change From Baseline in Maximum Inspiratory Pressure (MIP)
Description: Results for Cohorts 1, 2 and 3 are pooled as specified in the protocol.
Time Frame: Baseline, Week 12, Week 24, Week 36 and Week 48
Population: as for outcome 10
Measure: Mean (Standard Deviation); unit: cm H2O
Arm/Group | Cohorts 1, 2 and 3: SMT C1100
Number analyzed (Participants) | 36
cm H2O
  Week 12 Change from Baseline | 3.6 (32.68)
  Week 24 Change from Baseline: number analyzed (Participants) | 35
  Week 24 Change from Baseline | 3.0 (25.00)
  Week 36 Change from Baseline: number analyzed (Participants) | 31
  Week 36 Change from Baseline | 9.0 (18.40)
  Week 48 Change from Baseline: number analyzed (Participants) | 32
  Week 48 Change from Baseline | 8.7 (20.30)

13. Secondary Outcome: Change From Baseline in Maximum Expiratory Pressure (MEP)
Description: Results for Cohorts 1, 2 and 3 are pooled as specified in the protocol.
Time Frame: Baseline, Week 12, Week 24, Week 36 and Week 48
Population: as for outcome 10
Measure: Mean (Standard Deviation); unit: cm H2O
Arm/Group | Cohorts 1, 2 and 3: SMT C1100
Number analyzed (Participants) | 35
cm H2O
  Week 12 Change from Baseline | 1.8 (17.97)
  Week 24 Change from Baseline: number analyzed (Participants) | 34
  Week 24 Change from Baseline | 2.5 (22.95)
  Week 36 Change from Baseline: number analyzed (Participants) | 31
  Week 36 Change from Baseline | -1.0 (23.53)
  Week 48 Change from Baseline: number analyzed (Participants) | 31
  Week 48 Change from Baseline | 6.5 (20.09)

14. Secondary Outcome: Change From Baseline in Peak Expiratory Flow (PEF)
Description: Results for Cohorts 1, 2 and 3 are pooled as specified in the protocol.
Time Frame: Baseline, Week 12, Week 24, Week 36 and Week 48
Population: as for outcome 10
Measure: Mean (Standard Deviation); unit: Percentage of PEF
Arm/Group | Cohorts 1, 2 and 3: SMT C1100
Number analyzed (Participants) | 34
Percentage of PEF
  Week 12 Change from Baseline: number analyzed (Participants) | 32
  Week 12 Change from Baseline | 0.5 (20.65)
  Week 24 Change from Baseline | -0.1 (23.86)
  Week 36 Change from Baseline: number analyzed (Participants) | 32
  Week 36 Change from Baseline | -0.4 (23.46)
  Week 48 Change from Baseline: number analyzed (Participants) | 32
  Week 48 Change from Baseline | 9.6 (30.09)

15. Secondary Outcome: Change From Baseline in Peak Cough Flow (PCF)
Description: Analysis of PCF was planned for Cohort 3 only.
Time Frame: Baseline, Week 12, Week 24, Week 36 and Week 48
Population: No evaluable data was collected from Cohort 3 participants due to early study termination.
Arm/Group | Cohort 3: SMT C1100 Formulation 1
Number analyzed (Participants) | 0

16. Secondary Outcome: Change From Baseline in Sniff Nasal Inspiratory Pressure (SNIP)
Description: Analysis of SNIP was planned for Cohort 3 only.
Time Frame: Baseline, Week 12, Week 24, Week 36 and Week 48
Population: No evaluable data was collected from Cohort 3 participants due to early study termination.
Arm/Group | Cohort 3: SMT C1100 Formulation 1
Number analyzed (Participants) | 0

17. Secondary Outcome: Number of Participants That Experienced a Clinically Significant Change in Vital Signs Measurements
Description: Systolic blood pressure (SBP), diastolic blood pressure (DBP) and pulse will be disclosed with the following categories:
  * All values within 20% of change from baseline (< 20% change).
  * At least one value ≥ 20% reduction from baseline, but no increases ≥ 20% from baseline (≥ 20% reduction and no < 20% increase).
  * At least one value ≥ 20% increase from baseline, but no reductions ≥ 20% from baseline (≥ 20% Increase and no < 20% reduction).
  * At least one value ≥ 20% reduction from baseline and at least one value ≥ 20% increase from baseline (≥ 20% reduction and ≥ 20% increase).
  Results for Cohorts 1, 2 and 3 are pooled as specified in the protocol.
Time Frame: Baseline to Week 48
Population: as for outcome 10
Measure: Count of Participants; unit: Participants
Arm/Group | Cohorts 1, 2 and 3: SMT C1100
Number analyzed (Participants) | 40
Participants
  SBP: < 20% change | 28
  SBP: ≥ 20% reduction and no < 20% increase | 2
  SBP: ≥ 20% Increase and no < 20% reduction | 10
  SBP: ≥ 20% reduction and ≥ 20% increase | 0
  DBP: < 20% change | 19
  DBP: ≥ 20% reduction and no < 20% increase | 11
  DBP: ≥ 20% Increase and no < 20% reduction | 10
  DBP: ≥ 20% reduction and ≥ 20% increase | 0
  Pulse: < 20% change | 21
  Pulse: ≥ 20% reduction and no < 20% increase | 6
  Pulse: ≥ 20% Increase and no < 20% reduction | 13
  Pulse: ≥ 20% reduction and ≥ 20% increase | 0

18. Secondary Outcome: Number of Participants That Experienced a Clinically Significant in Physical Examination Result
Description: Examinations included: ear, nose and throat, cardiovascular system, pulmonary system, skin, abdomen, neurological system, height and weight. Results for Cohorts 1, 2 and 3 are pooled as specified in the protocol.
Time Frame: Day 1 to Week 48
Population: All participants who received at least one dose of study medication.
Measure: Count of Participants; unit: Participants
Arm/Group | Cohorts 1, 2 and 3: SMT C1100
Number analyzed (Participants) | 43
Participants | 1

19. Secondary Outcome: Number of Participants That Experienced a Potentially Clinically Significant Electrocardiogram Measurements
Description: PR interval (PRI), heart rate (HR), QTcF and increase from baseline in QTcF (IQTcF) were summarized categorically. Results for Cohorts 1, 2 and 3 are pooled as specified in the protocol.
Time Frame: Baseline to Week 48
Population: as for outcome 10
Measure: Count of Participants; unit: Participants
Arm/Group | Cohorts 1, 2 and 3: SMT C1100
Number analyzed (Participants) | 40
Participants
  PRI: <170 ms | 37
  PRI: ≥170 ms | 3
  PRI: < 20% change | 35
  PRI: ≥ 20% reduction and no < 20% increase | 2
  PRI: ≥ 20% increase and no < 20% reduction | 3
  PRI: ≥ 20% reduction and ≥ 20% increase | 0
  HR: < 20% change | 7
  HR: ≥ 20% reduction and no < 20% increase | 6
  HR: ≥ 20% increase and no < 20% reduction | 22
  HR: ≥ 20% reduction and ≥ 20% increase | 5
  QTcF: < 450 ms | 40
  QTcF: ≥ 450 ms | 0
  IQTcF: < 30 ms | 32
  IQTcF: 30 - 59 ms | 8
  IQTcF: >= 60 ms | 0

20. Secondary Outcome: Number of Participants That Experienced a Potentially Clinically Significant Echocardiogram Measurement
Description: Participants were at rest in a supine position for 10 minutes before the measurements were performed. Results for Cohorts 1, 2 and 3 are pooled as specified in the protocol.
Time Frame: Baseline, Week 24 and Week 48
Population: as for outcome 10
Measure: Count of Participants; unit: Participants
Arm/Group | Cohorts 1, 2 and 3: SMT C1100
Number analyzed (Participants) | 40
Participants
  Baseline: Normal | 38
  Baseline: Abnormal, Not Clinically Significant | 2
  Baseline: Abnormal, Clinically Significant | 0
  Week 24: number analyzed (Participants) | 38
  Week 24: Normal | 33
  Week 24: Abnormal, Not Clinically Significant | 5
  Week 24: Abnormal, Clinically Significant | 0
  Week 48: number analyzed (Participants) | 36
  Week 48: Normal | 33
  Week 48: Abnormal, Not Clinically Significant | 2
  Week 48: Abnormal, Clinically Significant | 1

21. Secondary Outcome: Number of Participants That Experienced a Clinically Significant Haematology Result (Investigator's Assessment)
Description: Parameters included: haemoglobin, haematocrit, mean corpuscular volume, white blood cells, red blood cells, neutrophils (percentage and absolute), lymphocytes (percentage and absolute), monocytes (percentage and absolute), eosinophils (percentage and absolute), basophils (percentage and absolute) and platelets. Results for Cohorts 1, 2 and 3 are pooled as specified in the protocol.
Time Frame: Day 1 to Week 48
Population: All participants who received at least one dose of study medication.
Measure: Count of Participants; unit: Participants
Arm/Group | Cohorts 1, 2 and 3: SMT C1100
Number analyzed (Participants) | 43
Participants | 0

22. Secondary Outcome: Number of Participants Who Experienced a Clinically Significant Biochemistry Result (Investigator's Assessment)
Description: Parameters included: calcium, potassium, sodium, albumin, urea nitrogen, uric acid, creatinine, creatine kinase, fasting glucose, cystatin C, lactate dehydrogenase, amylase, lipase, low density lipoprotein cholesterol, high density lipoprotein (HDL) cholesterol, cholesterol, non-HDL cholesterol, total HDL cholesterol ratio, total bilirubin, direct bilirubin, indirect bilirubin, alkaline phosphatase, alanine aminotransferase, aspartate aminotransferase, gamma glutamyl transferase and glutamate dehydrogenase. Results for Cohorts 1, 2 and 3 are pooled as specified in the protocol.
Time Frame: Day 1 to Week 48
Population: All participants who received at least one dose of study medication.
Measure: Count of Participants; unit: Participants
Arm/Group | Cohorts 1, 2 and 3: SMT C1100
Number analyzed (Participants) | 43
Participants | 3

23. Secondary Outcome: Number of Participants That Experienced a Potentially Clinically Significant Liver Function Result
Description: Laboratory measurements for alanine aminotransferase (ALT), aspartate aminotransferase (AST), total bilirubin (TB), alkaline phosphatase (ALP), and glutamate dehydrogenase (GLDH). Hy's Law is defined as an increase in ALT, AST and TB, indicating hepatocyte necrosis and functional deficit. Results for Cohorts 1, 2 and 3 are pooled as specified in the protocol.
Time Frame: Baseline to Week 48
Population: All participants who received at least one dose of study medication.
Measure: Count of Participants; unit: Participants
Arm/Group | Cohorts 1, 2 and 3: SMT C1100
Number analyzed (Participants) | 43
Participants
  ALT >= upper limit of normal (ULN) | 43
  ALT >= 2*ULN | 43
  ALT >= 3*ULN | 42
  AST >= ULN | 43
  AST >= 2*ULN | 42
  AST >= 3*ULN | 42
  TB >= ULN | 0
  TB >= 2*ULN | 0
  ALP >= 1.5*ULN | 0
  GLDH >= ULN excluding haemolysed samples | 27
  GLDH >= ULN including haemolysed samples | 30
  GLDH >= 2.5*ULN Excluding Haemolysed Samples | 2
  GLDH >= 2.5*ULN including haemolysed samples | 2
  Participants meeting Hy's law | 0

24. Secondary Outcome: Number of Participants That Experienced a Clinically Significant Urinalysis Result (Investigator's Assessment)
Description: Parameters included: glucose, bilirubin, ketones, specific gravity, blood, pH, protein, urobilinogen, nitrites and leucocytes. Results for Cohorts 1, 2 and 3 are pooled as specified in the protocol.
Time Frame: Day 1 to Week 48
Population: All participants who received at least one dose of study medication.
Measure: Count of Participants; unit: Participants
Groups:
- Cohort 1, 2 and 3: SMT C1100: Cohorts 1 and 3 participants received 2.5 g SMT C1100 formulation 1 orally twice-daily for at least 48 weeks. Cohort 2 participants received 1 g SMT C1100 formulation 2 orally twice-daily for at least 48 weeks.
Arm/Group | Cohort 1, 2 and 3: SMT C1100
Number analyzed (Participants) | 43
Participants | 0

25. Secondary Outcome: Number of Participants That Experienced a Clinically Significant Coagulation Result (Investigator's Assessment)
Description: Parameters included: activated partial thromboplastin time, prothrombin time and international normalised ratio. Coagulation was only assessed for Cohorts 2 and 3. Results for Cohorts 2 and 3 are pooled as specified in the protocol.
Time Frame: Day 1 to Week 48
Population: All participants who received at least one dose of study medication in Cohorts 2 and 3 only.
Measure: Count of Participants; unit: Participants
Groups:
- Cohorts 2 and 3 SMT C1100: Cohort 2 participants received 1 g SMT C1100 formulation 2 orally twice-daily for at least 48 weeks. Cohort 3 participants received 2.5 g SMT C1100 formulation 1 orally twice-daily for at least 48 weeks.
Arm/Group | Cohorts 2 and 3 SMT C1100
Number analyzed (Participants) | 13
Participants | 0

ADVERSE EVENTS:
Time Frame: Day 1 to a maximum of 96 weeks
Description: Treatment Emergent Adverse Events.
Arm/Group | Cohort 1: SMT C1100 Formulation 1 | Cohort 2: SMT C1100 Formulation 2 | Cohort 3: SMT C1100 Formulation 1
All-Cause Mortality (participants affected / at risk) | 0/30 | 0/10 | 0/3
Serious Adverse Events (participants affected / at risk) | 4/30 | 0/10 | 0/3
Other Adverse Events (participants affected / at risk) | 30/30 | 10/10 | 3/3
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Cohort 1: SMT C1100 Formulation 1 (N=30) | Cohort 2: SMT C1100 Formulation 2 (N=10) | Cohort 3: SMT C1100 Formulation 1 (N=3)
Femur fracture (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0)
Peripheral swelling (General disorders) | 1 (1) | 0 (0) | 0 (0)
Muscle spasms (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0)
Chromaturia (Renal and urinary disorders) | 1 (1) | 0 (0) | 0 (0)
Abdominal pain (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0)
Vomiting (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0)
Non-cardiac chest pain (General disorders) | 1 (1) | 0 (0) | 0 (0)
Viral infection (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Tonsillitis bacterial (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Rhabdomyolysis (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0)
Gastritis viral (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Spinal compression fracture (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Cohort 1: SMT C1100 Formulation 1 (N=30) | Cohort 2: SMT C1100 Formulation 2 (N=10) | Cohort 3: SMT C1100 Formulation 1 (N=3)
Faeces pale (Gastrointestinal disorders) | 18 | 3 | 3
Vomiting (Gastrointestinal disorders) | 17 | 6 | 0
Diarrhoea (Gastrointestinal disorders) | 12 | 4 | 2
Abdominal pain upper (Gastrointestinal disorders) | 8 | 3 | 1
Abdominal pain (Gastrointestinal disorders) | 7 | 0 | 0
Nausea (Gastrointestinal disorders) | 5 | 1 | 1
Constipation (Gastrointestinal disorders) | 2 | 1 | 1
Abdominal discomfort (Gastrointestinal disorders) | 2 | 1 | 0
Toothache (Gastrointestinal disorders) | 3 | 0 | 0
Faeces discoloured (Gastrointestinal disorders) | 1 | 1 | 0
Gastritis (Gastrointestinal disorders) | 2 | 0 | 0
Nasopharyngitis (Infections and infestations) | 6 | 5 | 0
Rhinitis (Infections and infestations) | 3 | 1 | 0
Upper respiratory tract infection (Infections and infestations) | 4 | 0 | 0
Ear infection (Infections and infestations) | 1 | 2 | 0
Gastroenteritis (Infections and infestations) | 2 | 1 | 0
Otitis media (Infections and infestations) | 3 | 0 | 0
Sinusitis (Infections and infestations) | 2 | 0 | 0
Viral upper respiratory tract infection (Infections and infestations) | 2 | 0 | 0
Campylobacter gastroenteritis (Infections and infestations) | 0 | 1 | 0
Gastroenteritis viral (Infections and infestations) | 0 | 1 | 0
Pharyngitis (Infections and infestations) | 0 | 1 | 0
Fall (Injury, poisoning and procedural complications) | 7 | 1 | 0
Procedural pain (Injury, poisoning and procedural complications) | 7 | 0 | 0
Contusion (Injury, poisoning and procedural complications) | 3 | 0 | 0
Head injury (Injury, poisoning and procedural complications) | 2 | 0 | 0
Joint injury (Injury, poisoning and procedural complications) | 2 | 0 | 0
Ligament sprain (Injury, poisoning and procedural complications) | 2 | 0 | 0
Skin abrasion (Injury, poisoning and procedural complications) | 2 | 0 | 0
Spinal fracture (Injury, poisoning and procedural complications) | 2 | 0 | 0
Foot fracture (Injury, poisoning and procedural complications) | 0 | 1 | 0
Pyrexia (General disorders) | 7 | 1 | 0
Fatigue (General disorders) | 4 | 1 | 0
Catheter site bruise (General disorders) | 2 | 0 | 0
Chest pain (General disorders) | 2 | 0 | 0
Cough (Respiratory, thoracic and mediastinal disorders) | 8 | 4 | 0
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 8 | 2 | 0
Rhinorrhoea (Respiratory, thoracic and mediastinal disorders) | 2 | 1 | 0
Sinus congestion (Respiratory, thoracic and mediastinal disorders) | 1 | 1 | 0
Wheezing (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0
Back pain (Musculoskeletal and connective tissue disorders) | 10 | 0 | 0
Pain in extremity (Musculoskeletal and connective tissue disorders) | 7 | 1 | 0
Arthralgia (Musculoskeletal and connective tissue disorders) | 3 | 1 | 1
Neck pain (Musculoskeletal and connective tissue disorders) | 2 | 0 | 0
Headache (Nervous system disorders) | 9 | 1 | 1
Dizziness (Nervous system disorders) | 0 | 1 | 0
Rash (Skin and subcutaneous tissue disorders) | 5 | 0 | 0
Swelling face (Skin and subcutaneous tissue disorders) | 3 | 0 | 0
Dry skin (Skin and subcutaneous tissue disorders) | 2 | 0 | 0
Erythema (Skin and subcutaneous tissue disorders) | 2 | 0 | 0
Pruritus (Skin and subcutaneous tissue disorders) | 2 | 0 | 0
Skin discolouration (Skin and subcutaneous tissue disorders) | 1 | 1 | 0
Aggression (Psychiatric disorders) | 2 | 1 | 0
Abnormal behaviour (Psychiatric disorders) | 1 | 1 | 0
Anger (Psychiatric disorders) | 0 | 1 | 1
Belligerence (Psychiatric disorders) | 0 | 1 | 0
Depressed mood (Psychiatric disorders) | 0 | 0 | 1
Enuresis (Psychiatric disorders) | 0 | 1 | 0
Irritability (Psychiatric disorders) | 0 | 1 | 0
Mood altered (Psychiatric disorders) | 0 | 1 | 0
Glutamate dehydrogenase increased (Investigations) | 3 | 1 | 0
Gamma-glutamyltransferase increased (Investigations) | 2 | 0 | 0
Decreased appetite (Metabolism and nutrition disorders) | 3 | 0 | 0
Increased appetite (Metabolism and nutrition disorders) | 1 | 1 | 0
Vitamin D deficiency (Metabolism and nutrition disorders) | 2 | 0 | 0
Vitreous floaters (Eye disorders) | 0 | 1 | 0
Skin papilloma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 3 | 0 | 0
Ear pain (Ear and labyrinth disorders) | 2 | 0 | 0
Cryptorchism (Congenital, familial and genetic disorders) | 0 | 1 | 0
Pollakiuria (Renal and urinary disorders) | 0 | 0 | 1
Dyspepsia (Gastrointestinal disorders) | 3 | 1 | 0
Lip swelling (Gastrointestinal disorders) | 3 | 0 | 0

LIMITATIONS AND CAVEATS:
Analysis of the data collected from Cohort 3 was limited as the study was terminated prior to the first participant's Week 24 visit.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes

DOCUMENTS (2):
  • Study Protocol (2017-02-24): https://cdn.clinicaltrials.gov/large-docs/62/NCT02858362/Prot_000.pdf
  • Statistical Analysis Plan (2018-04-05): https://cdn.clinicaltrials.gov/large-docs/62/NCT02858362/SAP_001.pdf